CLINICAL TRIAL: NCT03679234
Title: Impact of Infant Formula on Caregiver-perceived Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18.01.US.INF
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Healthy Infants

STUDY DESIGN:
Masking Description: Subjects and their parent/caregiver will be blinded to the intervention product. Care Providers at sites, Investigators, and Outcomes Assessors are unblinded to the intervention product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Routine infant formula
  Interventions: Other: Routine infant formula

INTERVENTIONS:
Other: Routine infant formula — Routine infant formula with probiotic

SUMMARY:
Understand the impact of switching to a commercially available infant formula on gastrointestinal symptoms

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant
* Full-term (> 37 weeks gestation)
* Birth weight > 2500 and < 4500 g
* 14-60 days of age on enrollment
* Singleton birth
* Infant's mother has elected not to breastfeed prior to enrollment
* Infant exclusively formula-fed for at least 5 days prior to enrollment
* Caregiver perceives infant as very or extremely fussy according to perceived fussiness based on the previous 3 days
* Caregiver wishes to switch infant's formula
* Has not received solid foods
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Known or suspected cow-milk allergy
* Currently receiving a specialty infant formula (e.g. thickened, extensively hydrolyzed, amino acid-based, metabolic)
* Has switched formula more than two times since hospital discharge
* Currently experiencing gastrointestinal or respiratory symptoms secondary to an ongoing infection or virus (e.g. gastrointestinal infection, upper respiratory infection, flu)
* Congenital illness or malformation that may affect infant feeding and/or growth
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrollment
* Receiving probiotic supplements
* Infant's family who in the Investigator's assessment cannot be expected to comply with treatment (feeding regimen).
* Participation in another study that has not been approved as a concomitant study by Nestlé Nutrition.

Ages: 14 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Infant GI Symptom Burden | 3 weeks
  Study personnel will administer questionnaire

SECONDARY OUTCOMES:
Formula Intake | 24 hours
  Caregivers will document on diary records
Fussiness | 24 hours
  Caregivers will document on diary records
Formula Satisfaction Questionnaire | 3 weeks
  Study personnel will administer questionnaire
Adverse Events | 24 hours and 3 weeks
  Assessed throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carvalho, MD, Study Director — Nestle Nutrition
Locations (7):
- United States (7):
  - Norwich Pediatrics Group, Norwich, Connecticut
  - Qualmedica Research, Owensboro, Kentucky
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Midsouth Center for Clinical Research, LLC, Memphis, Tennessee
  - ClinPoint Trials, Waxahachie, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No